CLINICAL TRIAL: NCT03393663
Title: Chronic Kidney Disease: Determinants of Progression and Cardiovascular Risk. A Cohort Study in a Brazilian Population
Brief Title: Chronic Kidney Disease: Determinants of Progression and Cardiovascular Risk
Acronym: PROGREDIR
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Silvia Maria de Oliveira Titan, Principal Investigator, MD-PhD, University of Sao Paulo
Other Study IDs: 2011/17341-0
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; cardiovascular disease; mortality; end stage renal disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine (midstream sample and 24h collection) and blood (fasting serum, fasting plasma, post OGGT serum, post OGGT plasma) aliquots were prepared and stored at -180 °C in nitrogen.
  DNA extraction was performed stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CKD-related outcomes — the study is observational

SUMMARY:
Chronic kidney disease has become an important Public Health issue in most developed and developing countries, with increasing incidence and prevalence rates. The cost associated with chronic kidney disease patients is very high, derived from renal replacement therapy and the cost associated with the high cardiovascular risk of this population. Primary and secondary preventive measures are imperative. In this sense, the comprehension of mechanisms and biomarkers associated with CKD progression and mortality risk in this population is an important area of research. Cohort studies are important tools for testing risk factors and biomarkers. Currently, CKD cohorts, particularly of those not on dialysis, are few and restricted to North America and Europe.

The present study established a cohort of 454 CKD participants (not on dialysis) in Sao Paulo, Brazil, who will be followed for 7-10 years. Baseline data collection was wide, including medical history, diet (food frequency questionnaire), calcium score, echocardiography, pulse wave velocity, cardiac frequency variability, carotid intimal media thickness, retinography, and an extensive biobank. Follow-up is ongoing and made through annual telephone interviews including questions on death, hospitalizations, and need of renal replacement therapy (RRT). Vital status is investigated periodically by a hot-pursuit strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the outpatient service of Hospital das Clínicas, São Paulo, Brazil.
* ≥ 30 years.
* at least two measurements of creatinine (with a minimum interval of 3 months) ≥ 1.6 mg/dl for men and ≥ 1.4 mg/ dl for women.

Exclusion Criteria:

* Patients attending oncology, psychiatry, human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS), viral hepatitis and glomerulonephritis services were excluded.
* hospitalization within the last six months;
* acute myocardial infarction within the last six months;
* autoimmune diseases;
* current pregnancy;
* psychiatric diseases;
* ongoing chemotherapy or immunosuppressive therapy;
* current renal replacement therapy;
* HIV/AIDS infection;
* hepatitis B or C;
* any organ transplantation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the outpatient service of Hospital das Clínicas, São Paulo, a public university facility providing quaternary-level care for patients with chronic diseases, were invited to participate in this study. Initially, from the outpatient records, all patients aged
  ≥ 30 years and at least two measurements of creatinine (with a minimum interval of 3 months) ≥ 1.6 mg/dl for men and ≥ 1.4 mg/ dl for women were considered potential candidates. Patients attending oncology, psychiatry, human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS), viral hepatitis and glomerulonephritis services were excluded. The remaining candidates were then contacted by phone and were invited to participate if they did not meet any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2013-12-15 (Actual); Study Completion 2013-12-15 (Actual)

PRIMARY OUTCOMES:
Overall Mortality | 7 years
  Mortality of any cause, confirmed by official death certificates obtained through several health offices (PRO-AIM, Fundação SEADE and National Mortality Registry).
Renal replacement therapy | 7 years
  Initiation of any modality of renal replacement therapy, even if not permanently.
  Besides participant information, RRT will be ascertained through the city and state´s Registries (Sao Paulo State Registry of Dialysis and Transplantation, Sao Paulo City Registry of Dialysis and Transplantation).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domingos MAM, Queiroz M, Lotufo PA, Bensenor IJ, Titan SMO. Serum RBP4 and CKD: Association with insulin resistance and lipids. J Diabetes Complications. 2017 Jul;31(7):1132-1138. doi: 10.1016/j.jdiacomp.2017.04.013. Epub 2017 Apr 18. PMID 28473187
- [Background] Domingos MA, Moreira SR, Gomez L, Goulart A, Lotufo PA, Bensenor I, Titan S. Urinary Retinol-Binding Protein: Relationship to Renal Function and Cardiovascular Risk Factors in Chronic Kidney Disease. PLoS One. 2016 Sep 21;11(9):e0162782. doi: 10.1371/journal.pone.0162782. eCollection 2016. PMID 27655369
- [Result] Domingos MAM, Goulart AC, Lotufo PA, Bensenor IJM, Titan SMO. Chronic kidney disease - determinants of progression and cardiovascular risk. PROGREDIR cohort study: design and methods. Sao Paulo Med J. 2017 Mar-Apr;135(2):133-139. doi: 10.1590/1516-3180.2016.0272261116. Epub 2017 Apr 20. PMID 28443950